CLINICAL TRIAL: NCT07349290
Title: Vitamin D (Bio)Fortified Shopping Baskets to Improve Vitamin D Status: a Household-level RCT
Brief Title: Vitamin D (Bio)Fortified Shopping Baskets to Improve Vitamin D Status
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Foodovation North West Regional College (Unknown); Kenedy Bacon (Unknown); Sofina Foods Europe (Unknown); Humanativ Ltd (Unknown); Agri-Food and Biosciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/24/0076
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Vitamin D Biofortification; Vitamin D Fortification; Vitamin D Status
Keywords: Vitamin D; Biofortification; Fortification; Household; Vitamin D Status
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Randomised unblinded parallel household trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (bio)fortified foods (Experimental)
  Interventions: Other: Vitamin D (bio)fortified food basket
- Control foods (Experimental)
  Interventions: Other: Control food basket

INTERVENTIONS:
Other: Vitamin D (bio)fortified food basket — Basket of vitamin D (bio)fortified foods provided to a household for consumption
  Arms: Vitamin D (bio)fortified foods
Other: Control food basket — Basket of control foods provided to a household for consumption
  Arms: Control foods

SUMMARY:
Vitamin D is essential for healthy bones, muscles, and immune function. It comes from food, supplements, and sunlight. There are two main forms; vitamin D2, found mainly in plant foods, and vitamin D3, which comes from animal foods and is more effective at increasing vitamin D levels in the body. In the UK, sunlight is often too weak especially in winter for the body to make enough vitamin D, so people rely mainly on dietary sources and supplements. Despite this, many people in the UK have low vitamin D levels, and teenagers are particularly at risk due to increased needs during growth, with around one in five adolescents having low vitamin D levels. Poor intake of vitamin D-rich foods, low supplement use, and inconsistent food fortification contribute to this problem. This study aims to assess whether a family-based household diet using natural and fortified vitamin D foods during winter can improve vitamin D levels in adolescents.

DETAILED DESCRIPTION:
Vitamin D is important for keeping bones, muscles, and the immune system healthy. There are two main types of vitamin D; vitamin D2, which mainly comes from plant-based foods, and vitamin D3, which mostly comes from animal foods and sunlight. Vitamin D3 is better at raising vitamin D levels in the body. After vitamin D is consumed or made in the skin, it is processed by the liver and kidneys into an active form that the body can use. People get vitamin D from food, supplements, and sunlight. Natural food sources include oily fish, meat, eggs, and liver. Some foods, such as breakfast cereals, spreads, and yoghurts, have vitamin D added to them (fortified foods). A small number of foods, like certain mushrooms, eggs, and bread, are also biofortified to contain higher levels of vitamin D. However, in countries like the UK, sunlight is often not strong enough especially in winter to allow the body to make enough vitamin D, so people rely more on food and supplements. Vitamin D levels are measured using a blood test. In the UK, a large proportion of the population has low vitamin D levels, with many people being either deficient or insufficient. Low vitamin D increases the risk of weak bones and bone diseases, such as rickets in children and osteoporosis in adults. Teenagers are especially at risk because their bodies need more vitamin D during periods of rapid growth. National surveys show that nearly one in five adolescents in the UK has low vitamin D levels, particularly during winter. Low intake of vitamin D-rich foods, limited supplement use, and reduced sunlight exposure all contribute to this problem. Although some foods in the UK are fortified with vitamin D, fortification is voluntary, meaning vitamin D levels vary widely between products. This makes it difficult for families to meet their vitamin D needs through diet alone. While studies have shown that vitamin D fortification can improve vitamin D levels, most research has focused on single foods rather than looking at the whole family diet. There is limited evidence on whether using a range of vitamin D-rich and fortified foods at home can help improve vitamin D levels in adolescents. This study aims to assess whether a family-based, household-level dietary intervention using natural and fortified vitamin D foods during winter can improve vitamin D status in families with adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Households with at least one adult member (≥18 years) and at least one adolescent member (11-17 years).
* Participants willing to consume the majority of study foods provided
* Participants willing to provide a total of two blood samples (maximum 25ml at each timepoint).

Exclusion Criteria:

* Any food allergies or intolerances, including anaphylaxis allergies
* Individuals taking/unwilling to stop taking high dose vitamin D supplements (1000 IU) for a washout period (4 weeks before) and for the duration of the study period
* Other major dietary exclusions, e.g. those following vegan or vegetarian lifestyles.
* Individuals with conditions causing malabsorption, e.g. coeliac disease

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Vitamin D status | From enrolment to the end of treatment at 4 weeks, comparison between treatments
  Measured by LC-MS/MS for 25(OH)D concentrations (µmol/L)

SECONDARY OUTCOMES:
Vitamin D intake | From enrolment to the end of treatment at 4 weeks, comparison between treatments
  Measured by validated Food Frequency Questionnaire, reported as average vitamin D intake µg/day.
Acceptability of food baskets | From enrolment to the end of treatment at 4 weeks, comparison between treatments
  Measured by qualitative interview to assess acceptability of food baskets provided to households
Knowledge of vitamin D | From enrolment to the end of treatment at 4 weeks, comparison between treatments
  Measured by quantitative (percentage score between 0% and 100%, higher score indicating better knowledge) and qualitative (open ended questions) questionnaire to assess knowledge of vitamin D
Perceptions and habits of vitamin D | From enrolment to the end of treatment at 4 weeks, comparison between treatments
  Measured by quantitative and qualitative (open ended questions) questionnaire to assess perception and habits of vitamin D

CONTACTS AND LOCATIONS:
Locations (1):
- Ulster University, Human Intervention Studies Unit, Coleraine, Co. Londonderry, Coleraine, United Kingdom

IPD SHARING:
Plan to Share IPD: No